CLINICAL TRIAL: NCT05045365
Title: A Prospective Study: Perfusion Assessment Using Blood Oxygen Level Dependent Functional Magnetic Resonance Angiographic Imaging and Parenchymal Blood Volume Imaging in Endovascular Treatment of Peripheral Arterial Occlusive Disease
Brief Title: Perfusion Assessment Using BOLD MRI and PBV in Endovascular Treatment of Peripheral Arterial Occlusive Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LBXZ-2105
Record Dates: First submitted 2021-06-02; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Peripheral Arterial Disease; Tissue Perfusion
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Current assessment of lower limb ischemia cannot reflect the location and degree of ischemia. Tissue perfusion assessment was used in the diagnosis and treatment of lower limb ischemia in this project, and the quantitative evaluation of ischemia degree was realized by using its advantages of quantitative analysis and perfusion imaging.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been diagnosed as PAOD by symptom and imaging;
* Subject intends to take endovascular treatment in PUMCH;
* Subjects without heavy stenosis in infrapopliteal artery (stenosis<30%), or with short length lesion(length≤5cm, stenosis≥30%);
* Age > 35 and < 80;
* Subject has been informed the study and has signed informed consent;

Exclusion Criteria:

* Subject with MRI contraindications or allergic to iodinated contrast medium;
* Subject underwent intervention therapy or angioplasty in target vessel within the last 3 months;
* Subject after stent implantation in superficial femoral artery;
* Subject with severe heart dysfunction, renal dysfunction, or cancer;

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study was conducted in PAOD patients aged 35 to 80 years with clinical symptoms such as claudication, resting pain, or ulceration, who were intended for endovascular treatment. Computed tomographic angiography disclosed the occlusive lesion in their target lesion. Subject with complex infrapopliteal lesions was excluded in order to reduce the influence of other variables.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Perfusion of the index leg assessed by BOLD MRI before and after endovascular intervention. | 1 year
  BOLD evaluates perfusion noninvasively and can be used for long-term monitoring and postoperative follow-up. Improving the perfusion assessment will improve the evaluation system for endovascular treatment of PAOD.
Perfusion of the index leg assessed by PBV before and after endovascular intervention. | During operation
  PBV can evaluate intraoperative perfusion quantitatively in real time.

SECONDARY OUTCOMES:
The relationship between perfusion and function of the lower limb in PAOD patients | 1 year
  The preoperative and postoperative motor functions of the patients were tested to analyze the functional impact of perfusion improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China